CLINICAL TRIAL: NCT04377139
Title: Observational, Epidemiological, Retrospective Study of the Management of CMV Infection in a Cohort of Patients Receiving Lung Transplantation in Spain
Brief Title: Management of Cytomegalovirus (CMV) Infection in Lung Transplant Recipients (LTR)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PR(AG)54/2020
Record Dates: First submitted 2020-05-03; First posted 2020-05-06 (Actual); Last update posted 2020-05-11 (Actual); Status verified 2020-05

CONDITIONS: Lung Transplant; Complications
Keywords: cytomegalovirus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Prophylaxis: Those LTR receiving prophylaxis against CMV
  Interventions: Procedure: Prophylaxis
- Preemptive therapy: Those LTR receiving preemptive therapy against CMV
  Interventions: Procedure: Preemptive

INTERVENTIONS:
Procedure: Prophylaxis — The intervention consists of analyzing the differences in the evolution of lung transplant recipients in relation to the intervention of prophylaxis or preemptive therapy against CMV in LTR
  Groups: Prophylaxis
Procedure: Preemptive — The intervention consists of analyzing the differences in the evolution of lung transplant recipients in relation to the intervention of prophylaxis or preemptive therapy against CMV in LTR
  Groups: Preemptive therapy

SUMMARY:
Background: Lung transplant recipients (LTR) have the highest risk of CMV infection. CMV pneumonitis, lymphocytic bronchitis, and detection of CMV DNA in bronchoalveolar lavage fluid are independent risk factors for the development of chronic lung allograft dysfunction (CLAD). However, to demonstrate the clinical impact of the indirect effects of CMV, it is necessary to conduct studies with a very large sample size.

Hypothesis: The different current preventive strategies for CMV infection in LTR and their clinical application on a daily basis impact on the development of direct and indirect effects of CMV in this population.

Objectives: To study the effect of CMV infection on LTR in relation to current preventive strategies in terms of:

* The incidence of acute and chronic rejection
* The incidence of other opportunistic infections
* The incidence of neoplastic disease, especially, post-transplant lymphoproliferative disease
* Patient and graft survival Methods: Multicenter, retrospective, cohort study. Consecutive inclusion of all adult lung transplant recipients from 2013 to 2017 with 2 years of follow-up. The investigators will collect and analyze the main clinical and microbiological variables in order to respond to the objectives of the study.

Relevance: Knowing in detail the current epidemiology of CMV infection in LTR and its subsequent influence on both mortality and the presence of different complications, could allow improving the management of these patients in the future.

ELIGIBILITY:
Inclusion Criteria:

· Survival > 1 month post-transplant

• High to moderate risk patients to develop CMV disease by means of pre-transplant CMV serology:

* Donor positive to recipient negative
* Recipient positive independently of donor serology

Exclusion Criteria:

* Survival < 1 month after procedure
* Low risk serology to develop CMV disease: both donor and recipient seronegative

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All those LTR performed in Spain during the study period
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
CMV infection and/or disease | Two-year follow-up
  Incidence

SECONDARY OUTCOMES:
Graft rejection both acute or CLAD | Two-year follow-up
  Incidence